CLINICAL TRIAL: NCT00192244
Title: A Prospective, Randomized, Double-Blind, Placebo-Controlled, Trial to Determine the Safety and Efficacy of Influenza Virus Vaccine, Trivalent, Types A & B, Live Cold-Adapted (CAIV-T) in Healthy Children
Brief Title: Trial to Determine the Safety and Efficacy of Influenza Virus Vaccine, Trivalent, Types A & B, Live, Cold-Adapted (CAIV-T) in Healthy Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: D153-P501
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2006-10-03 (Estimated); Status verified 2006-10

CONDITIONS: Healthy
MeSH Terms: interventions — Fluid Therapy

INTERVENTIONS:
Biological: CAIV-T, Liquid

SUMMARY:
- The purpose of this study is to determine the efficacy of CAIV-T in a diverse Asian population aged from 6 months to less than 36 months, in tropical and temperate climates, against culture-confirmed influenza illness. In addition, the trial provides the opportunity to investigate the efficacy of CAIV-T over multiple influenza seasons, and to investigate the effect of CAIV-T on acute otitis media.

ELIGIBILITY:
Inclusion Criteria:

* who are greater than or equal to 6 months and less than 36 months of age at the time of enrollment, and in good health as determined by medical history, physical examination, and clinical judgment;
* whose parent or legal guardian has provided written informed consent after the nature of the study has been explained;
* who, along with their parent or legal guardian, will be available for the duration of the study (24 months);
* whose parent/legal guardian can be reached by study staff for the post-immunization contacts [via telephone, clinic or home visits].

Exclusion Criteria:

* whose parents or caregiver are perceived to be unreliable or difficult to contact for evaluation or study visits during the study period;
* with any serious chronic disease (e.g., with signs of cardiac or renal failure or severe malnutrition), including progressive neurological disease;
* with Down's syndrome or other known cytogenetic disorders;
* with a known or suspected disease of the immune system or those receiving immunosuppressive therapy, including systemic corticosteroids;
* who received any blood products, including immunoglobulin, in the period from six months prior to vaccination through to the conclusion of the study;
* for whom there is intent to administer any other investigational vaccine or agent from one month prior to enrollment through to the conclusion of the study;
* with an immunosuppressed or compromised individual living in the same household;
* who, at any time prior to entry into this study, received a dose of any influenza vaccine (commercial or investigational);
* who were administered any live virus vaccine within one month prior to study vaccination or expected receipt of another live virus within one month of vaccination in this study;
* with a documented history of hypersensitivity to egg or egg protein, or any other component of the study vaccines or placebo;
* with a respiratory illness with wheezing within two weeks prior to enrollment;
* who received aspirin (acetylsalicylic acid) or aspirin-containing products in the two weeks prior to enrollment or for which use is anticipated during the study;
* with any medical conditions that in the opinion of the Investigator might interfere with interpretation of the study results; Note: A pregnant household member or day care provider is not considered a contraindication to enrollment.

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3000
Dates: Start 2000-09; Study Completion 2002-10

PRIMARY OUTCOMES:
The primary endpoint for efficacy is the first episode during the first year in a study child of a culture-confirmed influenza-illness, caused by community-acquired subtypes.

SECONDARY OUTCOMES:
The secondary endpoint for efficacy is the first episode during the second year in a study child of a culture-confirmed influenza-illness.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Walker, MD, Study Director — MedImmune LLC
Locations (1):
- The Prince of Wales Hospital, Hong Kong, China